CLINICAL TRIAL: NCT05600036
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ESK-001 in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of ESK-001 in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESK-001-006
Record Dates: First submitted 2022-10-12; First posted 2022-10-31 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- ESK-001 Dose Level 1 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- ESK-001 Dose Level 2 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- ESK-001 Dose Level 3 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- ESK-001 Dose Level 4 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- ESK-001 Dose Level 5 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- Placebo (Placebo Comparator): Placebo administered as an oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ESK-001 — Oral tablet
  Arms: ESK-001 Dose Level 1; ESK-001 Dose Level 2; ESK-001 Dose Level 3; ESK-001 Dose Level 4; ESK-001 Dose Level 5
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This study will consist of a 4 week screening period, 12 week treatment period, and a 4 week follow up period for a total of 20 weeks. Each participant will be randomized to receive ESK-001 or placebo daily for 12 weeks. An open label extension study will be available for those patients who complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Total body weight >40 kg (88 lb)
* Men and woman age 18-75
* Men and Women must use highly effective methods of contraception for the entirety of the study

Exclusion Criteria:

* History of malignancy within the last 5 years
* Positive for HIV, Hepatitis B or C
* History of tuberculosis
* Diagnosis of non-plaque psoriasis
* Patients with QTcF >450 msec (males) or >470 msec (females) at screening
* Live vaccines

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (38):
  - Investigator Site #1029, Birmingham, Alabama
  - Investigator Site # 1001, Phoenix, Arizona
  - Investigator Site #1023, Rogers, Arkansas
  - Investigator Site #1021, Encinitas, California
  - Investigator Site # 1008, Fremont, California
  - Investigator Site #1024, Los Angeles, California
  - Investigator Site # 1018, Los Angeles, California
  - Investigator Site #1016, San Diego, California
  - Investigator Site # 1007, Santa Monica, California
  - Investigator Site # 1002, Sherman Oaks, California
  - Investigator Site #1039, Brandon, Florida
  - Investigator Site #1013, Brandon, Florida
  - Investigator Site #1030, Fort Lauderdale, Florida
  - Investigator Site #1025, Hialeah, Florida
  - Investigator Site #1028, Miami, Florida
  - Investigator Site #1042, Tampa, Florida
  - Investigator Site #1035, Macon, Georgia
  - Investigator Site #1043, Sandy Springs, Georgia
  - Investigator Site # 1005, Rolling Meadows, Illinois
  - Investigator Site #1011, Indianapolis, Indiana
  - Investigator Site #1027, South Bend, Indiana
  - Investigator Site #1036, Overland Park, Kansas
  - Investigator Site #1034, Louisville, Kentucky
  - Investigator Site #1017, Owensboro, Kentucky
  - Investigator Site #1026, Rockville, Maryland
  - Investigator Site #1009, Bay City, Michigan
  - Investigator Site # 1010, Clarkston, Michigan
  - Investigator Site #1038, Warren, Michigan
  - Investigator Site #1031, New Brighton, Minnesota
  - Investigator Site #1014, Las Vegas, Nevada
  - Investigator Site #1037, Portsmouth, New Hampshire
  - Investigator Site #1033, Oklahoma City, Oklahoma
  - Investigator Site # 1019, Portland, Oregon
  - Investigator Site #1022, Philadelphia, Pennsylvania
  - Investigator Site #1012, Rapid City, South Dakota
  - Investigator Site # 1015, Houston, Texas
  - Investigator Site #1006, San Antonio, Texas
  - Investigator Site #1041, South Jordan, Utah
- Canada (10):
  - Investigator Site #2001, Edmonton, Alberta
  - Investigator Sie #2008, Surrey, British Columbia
  - Investigator Site #2003, Winnipeg, Manitoba
  - Investigator Site #2006, London, Ontario
  - Investigator Site #2004, Mississauga, Ontario
  - Investigator Site #2007, North Bay, Ontario
  - Investigator Site #2005, Oakville, Ontario
  - Investigator Site #2009, Toronto, Ontario
  - Investigator Site #2002, Waterloo, Ontario
  - Investigator Site #2010, Québec, Quebec
- Czechia (5):
  - Investigator Site #5515, Svitavy, Pardubice
  - Investigator Site #5507, Nový Jičín
  - Investigator Site #5514, Pardubice
  - Investigator Site #5506, Prague
  - Investigator Site #5505, Prague

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ESK-001 10mg QD: ESK-001 10mg tablet once a day
- ESK-001 20mg QD: ESK-001 20mg tablet once a day
- ESK-001 40mg QD: ESK-001 40mg tablet once a day
- ESK-001 20mg BID: ESK-001 20mg tablet twice a day
- ESK-001 40mg BID: ESK-001 40mg tablet twice a day
- Placebo: Placebo tablet
Period: Overall Study
Arm/Group | ESK-001 10mg QD | ESK-001 20mg QD | ESK-001 40mg QD | ESK-001 20mg BID | ESK-001 40mg BID | Placebo
Started | 36 | 36 | 39 | 40 | 39 | 38
Completed | 36 | 30 | 33 | 37 | 35 | 33
Not Completed | 0 | 6 | 6 | 3 | 4 | 5
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 3 | 5
Not completed — Discontinued Prior to Dosing Due to the Blood Sample Logistics | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject Can't Continue With Week 16 Visit | 0 | 1 | 0 | 0 | 0 | 0
Not completed — The Patient was Terminated From The Study Due to Sponsor Requirements | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESK-001 10mg QD | ESK-001 20mg QD | ESK-001 40mg QD | ESK-001 20mg BID | ESK-001 40mg BID | Placebo | Total
Number analyzed (Participants) | 36 | 36 | 39 | 40 | 39 | 38 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 37 | 35 | 33 | 35 | 206
  >=65 years | 3 | 3 | 2 | 5 | 6 | 3 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.7) | 43.9 (11.99) | 49.5 (10.45) | 47.7 (12.52) | 47.9 (14.17) | 49.1 (11.67) | 47.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 13 | 17 | 13 | 7 | 74
  Male | 24 | 24 | 26 | 23 | 26 | 31 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 14 | 13 | 7 | 11 | 13 | 65
  Not Hispanic or Latino | 29 | 21 | 26 | 33 | 28 | 24 | 161
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Asian | 1 | 2 | 2 | 2 | 2 | 4 | 13
  Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 2 | 0 | 0 | 3
  Black or African American | 4 | 0 | 1 | 1 | 1 | 3 | 10
  White | 30 | 31 | 33 | 34 | 33 | 27 | 188
  Other | 0 | 2 | 2 | 1 | 1 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Psoriasis Area and Severity Index (PASI-75) Between Doses of ESK-001 and Placebo
Description: Proportion of patients with moderate to severe psoriasis achieving ≥75% reduction in PASI score
Time Frame: 12 weeks
Population: All Randomized and Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | ESK-001 10mg QD | ESK-001 20mg QD | ESK-001 40mg QD | ESK-001 20mg BID | ESK-001 40mg BID | Placebo
Number analyzed (Participants) | 36 | 36 | 39 | 39 | 39 | 38
Percentage | 19.4 [8.2 to 36.0] | 33.3 [18.6 to 51.0] | 56.4 [39.6 to 72.2] | 56.4 [36.6 to 72.2] | 64.1 [47.2 to 78.8] | 0 [0.0 to 9.3]
Statistical Analysis 1: Comparison: ESK-001 10mg QD vs Placebo; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: ESK-001 20mg QD vs Placebo; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: ESK-001 40mg QD vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: ESK-001 20mg BID vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: ESK-001 40mg BID vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: To Assess the Safety and Tolerability of ESK-001 Dose in Moderate to Severe Psoriasis Patients
Description: Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). See Adverse Events section.
Time Frame: 12 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | ESK-001 Dose Level 1 | ESK-001 Dose Level 2 | ESK-001 Dose Level 3 | ESK-001 Dose Level 4 | ESK-001 Dose Level 5 | Placebo
Number analyzed (Participants) | 36 | 36 | 39 | 39 | 39 | 38
Participants | 19 | 14 | 19 | 18 | 25 | 15

3. Secondary Outcome: To Assess the Response Rate in Static Physician's Global Assessment (sPGA) Score
Description: Proportion of patients achieving an sPGA score of "0" ("cleared") or "1" ("minimal")
Time Frame: 12 weeks
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | ESK-001 10mg QD | ESK-001 20mg QD | ESK-001 40mg QD | ESK-001 20mg BID | ESK-001 40mg BID | Placebo
Number analyzed (Participants) | 36 | 36 | 39 | 39 | 39 | 38
Participants | 6 | 14 | 21 | 19 | 23 | 3

4. Secondary Outcome: To Characterize the Pharmacokinetics (PK) of ESK-001
Description: Plasma concentrations and PK parameters of ESK-001.
Time Frame: 14 weeks
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | ESK-001 10mg QD | ESK-001 20mg QD | ESK-001 40mg QD | ESK-001 20mg BID | ESK-001 40mg BID | Placebo
Number analyzed (Participants) | 36 | 36 | 39 | 39 | 39 | 38
ng/ml | 11.9 (12.4) | 33.0 (49.9) | 50.7 (44.8) | 63.9 (44.8) | 174.0 (125.0) | 2.9 (10.5)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from Screening through end of study (Week 16).
Arm/Group | ESK-001 10mg QD | ESK-001 20mg QD | ESK-001 40mg QD | ESK-001 20mg BID | ESK-001 40mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/39 | 0/39 | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/36 | 1/39 | 3/39 | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 8/36 | 4/36 | 11/39 | 18/39 | 18/39 | 9/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESK-001 10mg QD (N=36) | ESK-001 20mg QD (N=36) | ESK-001 40mg QD (N=39) | ESK-001 20mg BID (N=39) | ESK-001 40mg BID (N=39) | Placebo (N=38)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ESK-001 10mg QD (N=36) | ESK-001 20mg QD (N=36) | ESK-001 40mg QD (N=39) | ESK-001 20mg BID (N=39) | ESK-001 40mg BID (N=39) | Placebo (N=38)
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 2 | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 1 | 3 | 3
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3
Headache (Nervous system disorders) | 0 | 2 | 4 | 3 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish after the earlier of: publication of the final multicenter publication or 24 months after completion of the Study.

Investigator will provide to Sponsor a copy of any publication at least 60 days prior to submission. Sponsor may delete any confidential or proprietary information of Sponsor from the publication. Investigator will delay any publication an additional 90 days if requested to enable Sponsor to secure patent protection.

DOCUMENTS (2):
  • Study Protocol (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT05600036/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT05600036/SAP_001.pdf